CLINICAL TRIAL: NCT07111806
Title: Intravenous Tirofiban Versus Placebo After Delayed Thrombolysis (4.5-24h) in Acute Ischemic Stroke (PEARL-TIRO): A Multicenter, Double-Blind, Double-Dummy, Randomized Controlled Trial
Brief Title: Intravenous Tirofiban After Delayed Thrombolysis in Stroke
Acronym: PEARL-TIRO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEARL-TIRO
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; thrombolysis; Tirofiban
MeSH Terms: conditions — Ischemic Stroke | interventions — Tirofiban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban group (Experimental)
  Interventions: Drug: Tirofiban
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirofiban — Tirofiban is administered as a loading dose and continuous intravenous infusion as soon as possible after the randomization.
  Arms: Tirofiban group
Drug: Placebo — Matched placebo will be infused in a similar fashion.
  Arms: Placebo group

SUMMARY:
A multicenter, double-blind, double-dummy, randomized trial evaluating the efficacy and safety of intravenous tirofiban in acute ischemic stroke (AIS) patients without large/medium vessel occlusion, who presented 4.5-24 hours after onset and received intravenous thrombolysis (IVT).

DETAILED DESCRIPTION:
This study is a multicenter, double-blind, double-dummy, randomized clinical trial designed to evaluate the efficacy and safety of intravenous tirofiban in acute ischemic stroke (AIS) patients without large/medium vessel occlusion, who presented 4.5-24 hours after onset and received intravenous thrombolysis (IVT). The primary outcome is the proportion of patients with a 90-day modified Rankin scale (mRS) of 0-1.

Study intervention: (1) Participants in the intervention group will receive intravenous tirofiban as soon as possible after the randomization. (2) Participants in the control group will receive matched intravenous placebo in the same approach.

All participants will receive standard medical treatment.

A total of 852 participants are anticipated to be recruited for this study, with 426 participants in each group (1:1 ratio).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older;
2. Clinical diagnosed acute ischemic stroke (AIS) with last known well time of 4.5-24 hours;
3. Any of the following presentation of AIS:

1) Treated with IVT followed by no significant change in neurological function; 2) Treated with IVT followed by early neurological deterioration; 4. NIHSS score ≥4 before randomization; 5. Able to receive the designated study drug within 60 minutes after IVT; 6. Written informed consent is obtained from patients and/or their legal representatives.

Exclusion Criteria:

1. Intracranial or subarachnoid hemorrhage confirmed by cranial computed tomography (CT) or magnetic resonance imaging (MRI), or any intracranial hemorrhage history;
2. CTA/MRA/DSA showed occlusion of the internal carotid artery, middle cerebral artery M1 or M2 segment, anterior cerebral artery A1 segment, and vertebrobasilar artery;
3. Presence of any of the following unequivocal cardiac sources of embolism: chronic or paroxysmal atrial fibrillation, sick sinus syndrome, mitral stenosis, mechanical valve, endocarditis, intracardiac clot or vegetation, myocardial infarction within three months, dilated cardiomyopathy, left atrial spontaneous echo contrast, ejection fraction less than 30%;
4. Pre-stroke modified Rankin scale (mRS)≥2;
5. Renal insufficiency (glomerular filtration rate < 30 mL/min or serum creatinine > 220 μmol/L [2.5 mg/dl]);
6. Pregnant or lactating women;
7. NCCT, CTA source imaging, or MRI-DWI showing ASPECTS or PC-ASPECTS < 6;
8. Allergy to tirofiban, other glycoprotein IIb/IIIa inhibitors, aspirin or clopidogrel;
9. History of bleeding disorder, severe heart, liver or kidney disease, or sepsis;
10. Active bleeding diathesis, including clinical laboratory evidence of coagulation abnormalities (platelet count < 100×10⁹/L, activated partial thromboplastin time >50 seconds or international normalized ratio > 1.7), or treatment with a direct oral anticoagulant within the prior 48h;
11. CT or MR evidence of mass effect or intracranial tumor (except small meningioma);
12. CT or MR angiography evidence of intracranial arteriovenous malformations or aneurysm;
13. Severe allergy to contrast agents (non-mild rash allergy) or absolute contraindication to iodine contrast;
14. Any terminal illness with life expectancy less than 6 months;
15. Participating in other clinical trials;
16. Other conditions deemed unsuitable for the study by the investigator, such as inability to comprehend or comply with study procedures or follow-up due to mental illness, cognitive or emotional disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
The modified Rankin Scale score (mRS) 0-1 | 90 (±14) days
  The proportion of mRS score 0-1 at 90 (±14) days.

SECONDARY OUTCOMES:
Distribution of modified Rankin Scale score at 90 days | 90 (±14) days
  The shift analysis of the 90-day mRS with 5-6 merged at 90 (±14) days.
The modified Rankin Scale score 0-2 | 90 (±14) days
  The proportion of mRS score 0-2 at 90 (±14) days.
Early neurological improvement | 48 (±12) hours
  The proportion of patients with a ≥30% decrease in National Institute of Health stroke scale score from baseline.
Quality of life (EQ-5D-5L) | 90 (±14) days
  Health-related quality of life measured by EQ-5D-5L scale score at 90 (±14) days.

OTHER OUTCOMES:
SAFETY OUTCOME: Symptomatic intracranial hemorrhage | 48 (±12) hours
  Rate of symptomatic intracranial hemorrhage (sICH) within 48 hours from randomization (Heidelberg bleeding classification)
SAFETY OUTCOME: Any intracranial hemorrhage | 48 (±12) hours
  Rate of any intracranial hemorrhage within 48 hours from randomization
SAFETY OUTCOME: Major extracranial bleeding | 48 (±12) hours
  Rate of major extracranial bleeding within 48 hours from randomization (as defined by the Global Utilization of Streptokinase and Tissue-type Plasminogen Activator for Occluded Coronary Arteries, GUSTO criteria: moderate and severe bleeding)
SAFETY OUTCOME: Mortality | 90(±14) days
  All-cause mortality within 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available from Principal Investigators (Prof. Yamei Tang) upon reasonable request 6 months after the trial completion.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after the trial completion.
Access Criteria: The IPD will be available from Principal Investigators (Prof. Yamei Tang) upon reasonable request.